CLINICAL TRIAL: NCT03530995
Title: A 2-Part, Non-randomized, Open-label Study to Evaluate the Effect of Itraconazole, Rifampicin, Rabeprazole, and Omeprazole on the Pharmacokinetics of Belumosudil (KD025)
Brief Title: Drug-drug Interaction Between Belumosudil, Itraconazole, Rifampicin, Rabeprazole, and Omeprazole in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: KD025-107; 2018-000316-16 (EudraCT Number)
Record Dates: First submitted 2018-04-13; First posted 2018-05-21 (Actual); Results first posted 2021-09-13 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Drug-drug Interaction; Autoimmune Diseases; Fibrotic Disease
MeSH Terms: conditions — Autoimmune Diseases | interventions — belumosudil; Itraconazole; Rabeprazole; Rifampin; Omeprazole

STUDY DESIGN:
Intervention Model Description: Two-Part, Non-Randomised
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1, Period 1 (Experimental): Drug: Belumosudil. Subjects will receive belumosudil 200 mg single dose on Day 1
  Interventions: Drug: Belumosudil
- Part 1, Period 2 (Experimental): Drug: Itraconazole. Subjects will receive itraconazole 200 mg QD on Day 1 through Day 7.
  Drug: Belumosudil. Subjects will receive belumosudil 200 mg + itraconazole 200 mg QD on Day 8 Subjects will receive itraconazole 200 mg QD on Day 9
  Interventions: Drug: Belumosudil; Drug: Itraconazole
- Part 1, Period 3 (Experimental): Drug: Rabeprazole. Subjects will receive rabeprazole 20 mg BID on Day 1 through Day 3.
  Drug: Belumosudil. Subjects will receive belumosudil 200 mg + rabeprazole 20 mg QD on Day 4.
  Interventions: Drug: Belumosudil; Drug: Rabeprazole
- Part 1, Period 4 (Experimental): Drug: Rifampicin. Subjects will receive rifampicin 600 mg QD on Day 1 through Day 9.
  Drug: Belumosudil. Subjects will receive belumosudil 200 mg on Day 10.
  Interventions: Drug: Belumosudil; Drug: Rifampicin
- Part 2, Period 1 (Experimental): Drug: Belumosudil. Subjects will receive belumosudil 200 mg BID on Day 1.
  Interventions: Drug: Belumosudil
- Part 2, Period 2 (Experimental): Drug: Omeprazole. Subjects will receive omeprazole 20 mg QD on Day 1 through Day 3.
  Drug: Belumosudil. Subjects will receive belumosudil 200 mg BID + omeprazole 20 mg QD on Day 4.
  Interventions: Drug: Belumosudil; Drug: Omeprazole

INTERVENTIONS:
Drug: Belumosudil — Development candidate
  Other Names: Rezurock; SLx-2119
Drug: Itraconazole — Perpetrator drug
  Arms: Part 1, Period 2
Drug: Rabeprazole — Perpetrator drug
  Arms: Part 1, Period 3
Drug: Rifampicin — Perpetrator drug
  Arms: Part 1, Period 4
Drug: Omeprazole — Perpetrator drug
  Arms: Part 2, Period 2

SUMMARY:
This is a single-center, 2-part, non-randomized, open-label study of the drug-drug interactions of belumosudil (KD025) with itraconazole, rifampicin, rabeprazole, and omeprazole in healthy male subjects.

DETAILED DESCRIPTION:
Part 1:

The primary objective of Part 1 of this study is to determine the effect of itraconazole, rifampicin, and rabeprazole on the pharmacokinetics of once daily (QD) orally administered belumosudil in healthy male subjects. Part 1 consists of 4 periods.

In each study period, subjects will receive a single dose of belumosudil, in the fed state. Additionally, in order to assess the effects of inhibition and induction of CYP3A4 and the elevation of gastric pH on belumosudil exposure, subjects will receive multiple doses of perpetrator drugs in Periods 2 to 4; a strong CYP3A4 inhibitor, itraconazole, in Period 2; a proton pump inhibitor, rabeprazole, in Period 3; and a strong CYP3A4 inducer, rifampicin, in Period 4.

Subjects will receive a total of 4 single oral dosses of investigative product (IP), 200 mg belumosudil QD, in the fed state over 4 periods (each lasting 3 days with a minimum washout of 2, 8, and 4 days following completion of Periods 1, 2, and 3, respectively). Subjects also will receive 9 single oral doses of itraconazole 200 mg (QD over 9 days) in Period 2; 7 single oral doses of rabeprazole 20 mg (BID over 3 days followed by QD on 1 day) in Period 3; and 9 single doses of rifampicin 600 mg (QD over 9 days) in Period 4.

A follow-up visit will take place 3 to 5 days post-final discharge.

Part 2:

The primary objective of Part 2 of this study is to determine the effect of omeprazole on the PK of a single-day twice daily (BID; every 12 hours [Q12h]) dose of belumosudil administered orally, in healthy male subjects. Part 2 consists of 2 periods.

In Period 1, subjects will receive a single dose of belumosudil, in the fed state. In Period 2, in order to assess the effects of inhibition and induction of CYP3A4 and the elevation of gastric pH on belumosudil exposure, subjects will receive multiple doses of a proton pump inhibitor, omeprazole.

Subjects will receive a total of 4 single oral doses of IP (200 mg belumosudil, BID [Q12h] on 2 occasions) in the fed state over 2 periods (each lasting 3 days with a minimum washout of 2 days between dosing in Period 1 and the start of dosing with non-IP in Period 2). Subjects will also receive 4 single oral doses of omeprazole 20 mg (QD over 4 days) in Period 2.

A follow-up visit will take place 3 to 5 days post-final discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Age 18 to 55 years
3. Good state of health (mentally and physically) as indicated by a comprehensive clinical assessment (detailed medical history and a complete physical examination), electrocardiogram (ECG) and laboratory investigations (hematology, clinical chemistry, and urinalysis)
4. Body weight ≥50 kg
5. Body mass index of 18.0 to 32.0 kg/m^2 or, if outside the range, considered not clinically significant by the investigator
6. Must be willing and able to communicate and participate in the whole study
7. Must provide written informed consent
8. Must adhere to the contraception requirements

Exclusion Criteria:

1. Subjects who had previously participated in any other investigational study drug trial in which receipt of an IP occurred within 90 days prior to dosing. (Subjects who had previously received belumosudil in Part 1 at least 90 days prior to dosing in Part 2 were eligible to participate.)
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects with pregnant partners
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type)
6. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening and admission
7. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
8. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
9. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
10. Positive drugs of abuse test result at screening and admission
11. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
12. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <80 mL/min using the Cockcroft-Gault equation
13. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator
14. Subject has a history or presence of any of the following:

    * Active gastrointestinal disease requiring therapy
    * Hepatic disease and/or alanine aminotransaminase (ALT) or aspartate aminotransaminase (AST) > ULN
    * Renal disease and/or serum creatinine > ULN
    * Other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
15. Subjects with a history of cholecystectomy or gall stones
16. Subject has QT interval corrected using Fridericia's formula (QTcF) intervals >450 msec at screening or admission
17. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients; including intolerance to itraconazole, rabeprazole, and rifampicin
18. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
19. Donation or loss of greater than 400 mL of blood within the previous 3 months
20. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol) or herbal remedies in the 14 days before IP administration.
21. Failure to satisfy the investigator of fitness to participate for any other reason

Subjects Agreed to the Following Restrictions During the Duration of the Study:

1. No alcohol during the 24-hour period prior to screening and the 24-hour period prior to admission in Period 1, and 24 hours prior to commencing non-IP treatment in Part 1, Periods 2 to 4 and Part 2, Period 2, until discharge for each treatment period.
2. No food or drinks containing grapefruit or cranberry from 24 hours prior to admission in Period 1, and 24 hours prior to commencing non-IP treatment in Part 1 Periods 2 to 4 and Part 2 Period 2, until discharge for each treatment period.
3. No food or drinks containing caffeine or other xanthines from 24 hours prior to admission until discharge for each treatment period.
4. No food containing poppy seeds for 48 hours prior to screening and for 24 hours prior to admission until discharge for each treatment period.
5. No unaccustomed or strenuous exercise from the 72-hour period before the screening visit and then from 24 hours prior to admission until discharge for each treatment period.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences Ltd, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schueller O, Willson A, Singh N, Lohmer L, Alabanza A, Patel J. A Phase 1 Pharmacokinetic Drug Interaction Study of Belumosudil Coadministered With CYP3A4 Inhibitors and Inducers and Proton Pump Inhibitors. Clin Pharmacol Drug Dev. 2022 Jul;11(7):795-806. doi: 10.1002/cpdd.1082. Epub 2022 Mar 1. PMID 35230741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single centre, non-randomised, open label, two-part study. Part 1 of the study was a 4-period sequential dose study in healthy male subjects. The estimated duration from screening to discharge from the study was approximately 10 weeks. Part 2 of the study was a 2-period sequential dose study in healthy males. The estimated duration from screening to discharge from the study was approximately 7 weeks.
Groups:
- Part 1 Belumosudil (KD025) QD Dosing: Subjects received a single dose of belumosudil 200 mg on 4 separate occasions, and multiple single doses of itraconazole, rabeprazole and rifampicin, on separate occasions, for 9,4 and 9 consecutive days, respectively.
- Part 2 Belumosudil (KD025) BID Dosing: Subjects received a twice daily dose of belumosudil 200 mg on 2 separate occasions, and single doses of omeprazole for 4 consecutive days.
Period: Part 1 Period 1; Part 2 Period 1
Arm/Group | Part 1 Belumosudil (KD025) QD Dosing | Part 2 Belumosudil (KD025) BID Dosing
Started | 35 | 38
Completed | 35 | 38
Not Completed | 0 | 0
Period: Part 1 Period 2; Part 2 Period 2
Arm/Group | Part 1 Belumosudil (KD025) QD Dosing | Part 2 Belumosudil (KD025) BID Dosing
Started | 35 | 38
Completed | 35 | 38
Not Completed | 0 | 0
Period: Part 1 Period 3
Arm/Group | Part 1 Belumosudil (KD025) QD Dosing | Part 2 Belumosudil (KD025) BID Dosing
Started | 35 | 0 (Period 3 is not applicable to part 2 of the study.)
Completed | 32 | 0 (Period 3 is not applicable to part 2 of the study.)
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 1 | 0
Period: Part 1 Period 4
Arm/Group | Part 1 Belumosudil (KD025) QD Dosing | Part 2 Belumosudil (KD025) BID Dosing
Started | 32 | 0 (Period 4 is not applicable to part 2 of the study.)
Completed | 30 | 0 (Period 4 is not applicable to part 2 of the study.)
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects Part 1: KD025 QD Dosing: Period 1: 200 mg KD025 QD alone; Period 2: 200 mg KD025 QD with Itraconazole; Period 3: 200 mg KD025 QD with Rabeprazole; Period 4: 200 mg KD025 QD with Rifampicin
- All Subjects in Part 2: KD025 BID Dosing: Period 1: 200 mg KD025 BID alone; Period 2: 200 mg KD025 BID with Omeprazole
- Total: Total of all reporting groups
Arm/Group | All Subjects Part 1: KD025 QD Dosing | All Subjects in Part 2: KD025 BID Dosing | Total
Number analyzed (Participants) | 35 | 38 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (11.8) | 32.6 (10.6) | 34.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 35 | 38 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 28 | 35 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
BMI (body mass index) [Mean (Standard Deviation); unit: kg/m^2] | 26.81 (3.00) | 25.94 (3.36) | 26.36 (3.20)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Cmax of KD025 and KD025m2 in Part 1
Description: Maximum concentration (Cmax) of the parent drug, KD025, Metabolite 1 (KD025m1), and Metabolite 2 (KD025m2) for belumosudil alone, belumosudil + itraconazole, belumosudil + rabeprazole, and belumosudil + rifampicin at 0 to 48 hours post-dose
Time Frame: Pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12,24,36, and 48 hours post-dose
Population: Subject in Part 1 who received belumosudil alone, belumosudil with itraconazole, belumosudil with rabeprazole, and belumosudil with rifampicin. The number of subjects who participated in the study may differ from the number of subjects with an observation due to missing samples at critical timepoints or protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 1, Period 1: Belumosudil Alone: Belumosudil 200 mg single dose on Day 1
- Part 1, Period 2: Belumosudil + Itraconazole: Itraconazole 200 mg QD on Day 1 through Day 7; Belumosudil 200 mg + Itraconazole 200 mg QD on Day 8; Itraconazole 200 mg QD on Day 9
- Part 1, Period 3: Belumosudil + Rabeprazole: Rabeprazole 20 mg BID on Day 1 through Day 3; Belumosudil 200 mg + Rabeprazole 20 mg QD on Day 4
- Part 1, Period 4: Belumosudil + Rifampicin: Rifampicin 600 mg QD on Day 1-9; Belumosudil 200 mg on Day 10.
Arm/Group | Part 1, Period 1: Belumosudil Alone | Part 1, Period 2: Belumosudil + Itraconazole | Part 1, Period 3: Belumosudil + Rabeprazole | Part 1, Period 4: Belumosudil + Rifampicin
Number analyzed (Participants) | 35 | 35 | 32 | 29
ng/mL
  Parent Drug KD025 | 1770 (31.3) | 2130 (31.0) | 227 (58.4) | 712 (35)
  KD025m2: number analyzed (Participants) | 35 | 35 | 29 | 29
  KD025m2 | 337 (54.7) | 221 (60.8) | 23.5 (70.7) | 148 (57.3)

2. Primary Outcome: Pharmacokinetics: Cmax of KD025m1 in Part 1
Description: Maximum concentration (Cmax) of Metabolite 1 (KD025m1) for belumosudil alone and for belumosudil + rifampicin up to 48 hours post-dose
Time Frame: Pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12,24,36, and 48 hours post-dose
Population: Subjects in Part 1 who received belumosudil alone and belumosudil with rifampicin. The number of subjects who participated in the study may differ from the number of subjects with an observation due to missing samples at critical timepoints or protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1, Period 1: Belumosudil Alone | Part 1, Period 4: Belumosudil + Rifampicin
Number analyzed (Participants) | 35 | 29
ng/mL | 23.2 (40.0) | 52.5 (34.0)

3. Primary Outcome: Pharmacokinetics: Cmax of KD025, KD025m1, and KD025m2 in Part 2
Description: Maximum concentration (Cmax) of the parent drug (KD025), for Metabolite 1 (KD025m1), and for Metabolite 2 (KD025m2), for belumosudil alone and for belumosudil + omeprazole up to 48 hours post-dose
Time Frame: Pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12,12.5,13,13.5,14,15,16,17,18,20,22,24,36, and 48 hours post-dose
Population: Subjects in Part 2 who received belumosudil alone and belumosudil with omeprazole. The number of subjects who participated in the study may differ from the number of subjects with an observation due to missing samples at critical timepoints or protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 2, Period 1: Belumosudil Alone: Belumosudil 200 mg BID (Q12h) on Day 1
- Part 2, Period 2: Belumosudil + Omeprazole: Omeprazole 20 mg QD fasted for 3 days (Period 2 Days -3 to -1), Omeprazole 20 mg QD fasted + Belumosudil 200 mg BID (Q12h) fed on 4th day (Period 2 Day 1)
Arm/Group | Part 2, Period 1: Belumosudil Alone | Part 2, Period 2: Belumosudil + Omeprazole
Number analyzed (Participants) | 38 | 38
ng/mL
  Cmax--1st dose: KD025: number analyzed (Participants) | 37 | 38
  Cmax--1st dose: KD025 | 1790 (34.5) | 575 (145.7)
  Cmax--2nd dose: KD025: number analyzed (Participants) | 38 | 37
  Cmax--2nd dose: KD025 | 1760 (37.0) | 903 (63.8)
  Cmax--1st Dose: KD025m1: number analyzed (Participants) | 36 | 19
  Cmax--1st Dose: KD025m1 | 23.8 (39.6) | 18.0 (54.6)
  Cmax--2nd Dose: KD025m1: number analyzed (Participants) | 36 | 20
  Cmax--2nd Dose: KD025m1 | 23.6 (46.4) | 18.9 (48.7)
  Cmax--1st Dose: KD025m2: number analyzed (Participants) | 37 | 35
  Cmax--1st Dose: KD025m2 | 282 (75.6) | 72.3 (166.8)
  Cmax--2nd Dose: KD025m2: number analyzed (Participants) | 38 | 36
  Cmax--2nd Dose: KD025m2 | 257 (83.9) | 115 (121.8)

4. Primary Outcome: Pharmacokinetics: AUC(0-inf) and AUC(0-24) of KD025 and KD025 m2 for Subject in Part 1 and Part 2
Description: Area under concentration-time curve from zero hours to infinity (AUC[0-inf]) and from zero hours to 24 hours post-dose (AUC[0-24)) for the parent drug KD025, and Metabolite 2, KD025m2, for subjects up to 48 hours each for Part 1 and for Part 2
Time Frame: Part 1: Pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12,24,36, and 48 hours post-dose; Part 2: Pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12,12.5,13,13.5,14,15,16,17,18,20,22,24,36, and 48 hours post-dose
Population: Subjects in Part 1 who received belumosudil alone, belumosudil with itraconazole, belumosudil with rabeprazole, and belumosudil with rifampicin; Subjects in Part 2 who received belumosudil alone and belumosudil with omeprazole. The number of subjects who participated in the study may differ from the number of subjects with an observation due to missing samples at critical timepoints or protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h)/mL
Groups:
- Part 1, Period 2: Belumosudil + Itraconazole: Itraconazole 200 mg QD on Day 1-7; Belumosudil 200 mg + Itraconazole 200 mg QD on Day 8; Itraconazole 200 mg QD on Day 9
- Part 1, Period 3: Belumosudil + Rabeprazole: Rabeprazole 20 mg BID on Day 1-3; Belumosudil 200 mg + Rabeprazole 20 mg QD on Day 4.
- Part 2, Period 1: Belumosudil Only: Belumosudil 200 mg BID (Q12h) fed on a single day, Period 1 Day 1
- Part 2, Period 2: Belumosudil + Omeprazole: Omeprazole 20 mg QD fasted for 3 days (Period 2, Days -3 to -1); Omeprazole 20 mg QD fasted + Belumosudil 200 mg BID (Q12h) fed on 4th day (Period 2 Day 1)
Arm/Group | Part 1, Period 1: Belumosudil Alone | Part 1, Period 2: Belumosudil + Itraconazole | Part 1, Period 3: Belumosudil + Rabeprazole | Part 1, Period 4: Belumosudil + Rifampicin | Part 2, Period 1: Belumosudil Only | Part 2, Period 2: Belumosudil + Omeprazole
Number analyzed (Participants) | 35 | 35 | 32 | 29 | 38 | 38
(ng*h)/mL
  AUC(0-inf): KD025: number analyzed (Participants) | 34 | 33 | 28 | 29 | 34 | 32
  AUC(0-inf): KD025 | 9080 (33.3) | 11200 (38.1) | 1680 (65.8) | 2500 (34.5) | 18800 (37.1) | 9880 (59.2)
  AUC(0-inf): KD025m2: number analyzed (Participants) | 28 | 29 | 2 | 23 | 29 | 15
  AUC(0-inf): KD025m2 | 1230 (69.5) | 843 (73.7) | 174 (11.1) | 396 (50.2) | 1900 (90.4) | 1110 (30.3)
  AUC(0-24): KD025: number analyzed (Participants) | 35 | 35 | 32 | 29 | 37 | 37
  AUC(0-24): KD025 | 8430 (30.5) | 10400 (35.8) | 1510 (60.7) | 2490 (34.1) | 16800 (36.4) | 7970 (58.9)
  AUC(0-24): KD025m2: number analyzed (Participants) | 35 | 35 | 21 | 29 | 37 | 37
  AUC(0-24): KD025m2 | 1100 (63.7) | 745 (70.7) | 110 (84.0) | 376 (56.7) | 1950 (82.3) | 767 (115.3)

5. Primary Outcome: Pharmacokinetics: AUC(0-24) of KD025m1 for Part 1 and for Part 2
Description: Area under concentration-time curve from zero hours to 24 hours post-dose (AUC[0-24]) for Metabolite 1, KD025m1, for subjects in Part 1 and for subjects in Part 2
Time Frame: Part 1: Pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12, and 24 hours post-dose; Part 2: Pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12,12.5,13,13.5,14,15,16,17,18,20,22, and 24 hours post-dose
Population: Subjects in Part 1 who received belumosudil alone and belumosudil with rifampicin; Subjects in Part 2 who received belumosudil alone and belumosudil with omeprazole. The number of subjects who participated in the study may differ from the number of subjects with an observation due to missing samples at critical timepoints or protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h)/mL
Groups:
- Part 2, Period 1: Belumosudil Alone: Belumosudil 200 mg BID (Q12h) fed on a single day, Period 1 Day 1
Arm/Group | Part 1, Period 1: Belumosudil Alone | Part 1, Period 4: Belumosudil + Rifampicin | Part 2, Period 1: Belumosudil Alone | Part 2, Period 2: Belumosudil + Omeprazole
Number analyzed (Participants) | 27 | 29 | 35 | 15
(ng*h)/mL | 75.6 (42.1) | 148 (41.9) | 138 (91.3) | 91.5 (76.3)

ADVERSE EVENTS:
Time Frame: Part 1, Period 1: 1 day Part 1, Period 2: 9 days Part 1, Period 3: 4 days Part 1, Period 4: 10 days Part 2, Period 1: 1 day Part 2, Period 2: 4 days
Groups:
- Part 1, Period 1: Belumosudil Only: Belumosudil 200 mg single dose on Day 1
- Part 1, Period 2: Belumosudil + Itraconazole: Itraconazole 200 mg QD Day 1-7, Belumosudil 200 mg QD with itraconazole on Day 8, Itraconazole 200 mg QD on Day 9
- Part 1, Period 3: Belumosudil +Rabeprazole: Rabeprazole 20 mg BID on Day 1-3, Belumosudil 200 mg + rabeprazole 20 mg QD on Day 4
- Part 1, Period 4: Belumosudil + Rifampicin: Rifampicin 600 mg QD on Day 1-9, Belumosudil 200 mg on Day 10
- Part 2, Period 1: Belumosudil Only: Belumosudil 200 mg BID (Q12h) fed on a single day, Period 1 Day 1: KD025 200 mg BID
- Part 2, Period 2: Belumosudil + Omeprazole: Omeprazole 20 mg QD fasted for 3 days (Period 2 Days -3 to -10, Omeprazole 20 mg QD fasted + Belumosudil 200 mg BID (Q12h) fed on 4th day (Period 2 Day 1)
Arm/Group | Part 1, Period 1: Belumosudil Only | Part 1, Period 2: Belumosudil + Itraconazole | Part 1, Period 3: Belumosudil +Rabeprazole | Part 1, Period 4: Belumosudil + Rifampicin | Part 2, Period 1: Belumosudil Only | Part 2, Period 2: Belumosudil + Omeprazole
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/33 | 0/32 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/35 | 0/33 | 0/32 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 6/35 | 9/35 | 6/33 | 8/32 | 9/38 | 5/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Period 1: Belumosudil Only (N=35) | Part 1, Period 2: Belumosudil + Itraconazole (N=35) | Part 1, Period 3: Belumosudil +Rabeprazole (N=33) | Part 1, Period 4: Belumosudil + Rifampicin (N=32) | Part 2, Period 1: Belumosudil Only (N=38) | Part 2, Period 2: Belumosudil + Omeprazole (N=38)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Period 1: Belumosudil Only (N=35) | Part 1, Period 2: Belumosudil + Itraconazole (N=35) | Part 1, Period 3: Belumosudil +Rabeprazole (N=33) | Part 1, Period 4: Belumosudil + Rifampicin (N=32) | Part 2, Period 1: Belumosudil Only (N=38) | Part 2, Period 2: Belumosudil + Omeprazole (N=38)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 6 (6) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Medical device site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding results. The sponsor cannot require changes to the study results in the communication except to remove sponsor's confidential information. Sponsor cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT03530995/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT03530995/SAP_001.pdf